CLINICAL TRIAL: NCT06735105
Title: Comparative Study on the Value of Three DWI Scan Sequences of 3.0T Magnetic Resonance in Staging of Gastric Cancer
Brief Title: Study on the Value of Three DWI Scanning Sequences in Staging of Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KYLX2023-167
Record Dates: First submitted 2024-11-27; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SS-EPI-DWI T-stage of gastric cancer (No Intervention)
- TSE-DWI T-stage of gastric cancer (Other)
  Interventions: Diagnostic Test: Scanning parameter
- ZOOM-DWI T-stage of gastric cancer (Other)
  Interventions: Diagnostic Test: Scanning parameter

INTERVENTIONS:
Diagnostic Test: Scanning parameter — Based on abdominal scanning, TSE-DWI,ZOOMIT DWI and EPI-DWI scans were performed, and the study was divided into two steps according to the nanomotion criteria. The first step was self-controlled, which was divided into experimental group and control group. The experimental group included TSE-DWI,ZOOMit DWI, and the control group included EPI-DWI. Then the image quality was evaluated by subjective and objective evaluation indexes. In the second step, the three DWI stages were performed separately by four diagnosticians, with an interval of 1 month, and statistical analysis was performed at the end.
  Arms: TSE-DWI T-stage of gastric cancer; ZOOM-DWI T-stage of gastric cancer

SUMMARY:
Accurate staging is critical for effective gastric cancer treatment planning. Conventional DWI (C-DWI) has limitations in image quality due to magnetic field inhomogeneity, which hampers precise T staging.

This study aims to compare the image quality and T staging accuracy of C-DWI, TSE-DWI, and ZOOMit-DWI (Z-DWI) sequences in MRI examinations of gastric cancer patients.

A prospective study plan to enroll 72 gastric cancer patients undergoing preoperative MRI with C-DWI, TSE-DWI, and Z-DWI sequences using a 3.0 T scanner. Quantitative metrics (ADC, SNR, CNR) and image quality were evaluated. T staging accuracy was assessed by comparing MRI results with postoperative pathological staging using ROC analysis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was diagnosed with gastric cancer by pathological biopsy
2. No biopsy was taken within 1 week before MR Examination to rule out the effect of bleeding on the image
3. No contraindications for MRI examination; And exclude serious heart, liver, kidney, cerebrovascular diseases.

Exclusion Criteria:

1. The image quality cannot meet the diagnostic criteria;
2. Patients could not tolerate MRI examination, resulting in incomplete MR-related sequence image data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
T staging of gastric cancer | one year
  Study on the value of three DWI scanning sequences in T staging of gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, China

IPD SHARING:
Plan to Share IPD: No